CLINICAL TRIAL: NCT04647188
Title: Measuring the Quality of Surgical Care and Setting Benchmarks for Training Using Intuitive Data Recorder Technology
Acronym: MASTERY
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Birmingham (Other)
Collaborators: Newcastle-upon-Tyne Hospitals NHS Trust (Other); Imperial College Healthcare NHS Trust (Other); Barts & The London NHS Trust (Other); Portsmouth Hospitals NHS Trust (Other Government); Royal Marsden NHS Foundation Trust (Other); Wirral University Teaching Hospital NHS Trust (Other); The Leeds Teaching Hospitals NHS Trust (Other); Guy's and St Thomas' NHS Foundation Trust (Other); South Tees Hospitals NHS Foundation Trust (Other); University Hospitals Coventry and Warwickshire NHS Trust (Other); Intuitive Surgical (Industry); University Hospitals, Leicester (Other); Sheffield Teaching Hospitals NHS Foundation Trust (Other); Golden Jubilee National Hospital (Other Government); Royal Surrey County Hospital NHS Foundation Trust (Other); Oxford University Hospitals NHS Trust (Other); The Christie NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: RG_19-041
Record Dates: First submitted 2020-10-08; First posted 2020-11-30 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-05

CONDITIONS: Cancer; Surgery
Keywords: Robotic assisted surgery (RAS)
MeSH Terms: conditions — Neoplasms | interventions — Robotic Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Urology group: Includes patients undergoing prostatectomy (n=100)
  Interventions: Other: Robotic assisted surgery with IDR data capture
- Colorectal group: Includes patients undergoing anterior rectal resection (n=100)
  Interventions: Other: Robotic assisted surgery with IDR data capture
- Thoracic group: Includes patients undergoing lobectomy or segmentectomy (n=100)
  Interventions: Other: Robotic assisted surgery with IDR data capture
- Gynaecological group: Includes patients undergoing hysterectomy (n=100)
  Interventions: Other: Robotic assisted surgery with IDR data capture
- HpB group: Includes pancreatic tumour resection patients (n=50)
  Interventions: Other: Robotic assisted surgery with IDR data capture
- Ear, Nose & Throat group: Includes patients undergoing lateral oropharyngectomy (n=50)
  Interventions: Other: Robotic assisted surgery with IDR data capture

INTERVENTIONS:
Other: Robotic assisted surgery with IDR data capture — Robotic assisted surgery with digital point of care data capture using Intuitive Data Recorder (IDR) technology

SUMMARY:
MASTERY is a multi-centre prospective cohort study involving patients undergoing robotic assisted surgery for prostate, colorectal, lung, gynaecological, hepatobiliary, and ear, nose & throat tumours.

DETAILED DESCRIPTION:
MASTERY will create a data collection platform to capture, annotate and analyse digital point of care data relating to surgeon's performance during live surgery. This is a multi-centre prospective cohort study involving patients undergoing robotic assisted surgery for prostate, colorectal, lung, gynaecological, hepatobiliary, and ear, nose & throat tumours. In this study, automated digital point of care data relating to the surgeons' performance will be collected via the Intuitive Data Recorder (IDR) device (Intuitive Surgical Inc, USA). Data collection will also encompass surgeon characteristics, patient characteristics, 30-day clinical outcomes including surgical complications, reoperation, length of stay and hospital readmission. This will also include collection of baseline, 30- and 90-day patient reported outcomes data.

MASTERY is the first study of the RCS Robotics Working Group and aims to initially recruit 500 patients across 13 centres in United Kingdom from January 2021.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 16years
* Patients undergoing robotic assisted surgery for prostate, colorectal, lung, gynaecological, hepatobiliary, and ENT tumours
* Patients consenting to data collection who are scheduled to undergo robotic assisted surgery

Exclusion Criteria:

* Age < 16years
* Patients undergoing robotic surgery for other indications not relevant to the study
* Patients not consenting to data capture

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will include patients undergoing robotic assisted surgery for .prostate, colorectal, lung, gynaecological, hepatobiliary, and ear, nose and throat tumours
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-03-09 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with surgical complication | Day 30 after surgery
  Surgical complication rate at day-30

OTHER OUTCOMES:
Total operating time per surgery | During the surgery
  Intraoperative outcome - total operating time in hours
Number of patients with blood loss greater than 500mls during surgery | During the surgery
  Intraoperative outcome - total blood loss
Number of patients with adverse events reported at day 30 | Day 30 after surgery
  Adverse events rate
Total hospital length of stay at day 30 | Day 30 after surgery
  Hospital length of stay
Number of patients with readmission at day 30 | Day 30 after surgery
  Readmission rate
Time to complete cardinal steps in minutes | During the surgery
  Time taken by surgeon to complete each surgery cardinal step
Number of patients with complete or incomplete surgical resection | During the surgery
  Intraoperative outcome - completeness of surgical resection (defined by the surgeon as "complete" or "incomplete")
Oncological parameter - tumour stage | Baseline
  Tumour stage defined by the TNM staging system
Number of robotic assisted surgeries carried out by surgeon prior to enrollment in study | Baseline
  Surgeon's caseload prior surgery
Patient reported outcomes | Baseline, day 30 and day 90 after surgery
  Patient's global assessment of quality of life via the EORTC QLQ-C30 and the specialty specific modules (PR25, LC29, EN24, CR29, H&N43)
  All of the scales and single-item measures range in score from 0 to 100. A high score for the Sexual Activity and Sexual Functioning scales represents a high level of functioning, whereas a high score for the Urinary, Bowel, and Hormonal Treatment-Related symptoms scales and Incontinence Aid item represents a high level of symptomatology or problems.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Bach, Principal Investigator — University of Birmingham; Royal College of Surgeons UK Robotics Group; Naeem Soomro, Principal Investigator — Newcastle-Upon-Tyne Hospitals NHS Trust; Royal College of Surgeons UK Robotics Group
Locations (15):
- United Kingdom (15):
  - University Hospitals Coventry & Warwickshire NHS Trust, Coventry
  - Golden Jubilee National Hospital, Glasgow
  - Royal Surrey NHS Foundation Trust, Guildford
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - Barts Health NHS Trust, London
  - Guy's and St Thomas' NHS Foundation Trust, London
  - The Royal Marsden Hospital, London
  - The Royal Marsden NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester
  - Wirral University Teaching Hospital NHS Foundation Trust, Metropolitan Borough of Wirral
  - South Tees NHS Foundation Trust, Middlesbrough
  - Newcastle Hospitals NHS Foundation Trust, Newcastle upon Tyne
  - Oxford University Hospitals NHS Foundation Trust, Oxford
  - Portsmouth Hospitals NHS Trust, UK, Portsmouth
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield

IPD SHARING:
Plan to Share IPD: No